CLINICAL TRIAL: NCT02658747
Title: A Retrospective Chart Review to Describe the Rate of Neutropenic Sepsis in Patients With Non-Small Cell Lung Cancer Treated With Single-Agent Docetaxel and Associated Resource Use in the UK
Brief Title: Neutropenic Sepsis in Patients With Non-Small Cell Lung Cancer Treated With Single-Agent Docetaxel and Associated Resource Use in the UK
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30033
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort Docetaxel: Participants initiated on docetaxel for the treatment of relapsed non-small cell lung cancer (NSCLC)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
This is a multi-center retrospective observational research study collecting data for participants initiated on docetaxel for the treatment of relapsed non-small cell lung cancer (NSCLC) up to 6 years before start of data collection and who have completed/stopped docetaxel treatment at least 30 days prior to data collection. The primary goal of this study is to describe the percentage of participants with at least one neutropenic sepsis (NS) episode following initiation of treatment with single-agent docetaxel. Data will be collected until end of docetaxel treatment plus an additional 30 days to allow for presentation with toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with locally advanced or metastatic (stage Ill or IV) non-small cell lung cancer (NSCLC)
* Relapsed disease following, or unable to tolerate, at least one line of prior chemotherapy
* Initiated on single-agent docetaxel up to a maximum of 6 years prior to date of collection
* Aged 18 years at date of first docetaxel dose
* Completed or stopped treatment with docetaxel at least 30 days prior to date of data collection

Exclusion Criteria:

* Receiving docetaxel in an interventional clinical trial
* For whom no details of absolute neutrophil count are recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants initiated on docetaxel for the treatment of relapsed non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Receiving Single-Agent Docetaxel Chemotherapy for Treatment of Relapsed Non-Small Cell Lung Cancer (NSCLC) with an Episode of Neutropenic Sepsis (NS) with an Absolute Neutrophil Count of Less Than 1.0 x 10^9/L | Up to 6 years

SECONDARY OUTCOMES:
Frequency with which Participants Attend Hospital for Management of Specified Hematological Docetaxel-Related Toxicities, Including Anemia, Thrombocytopenia, Neutropenia, Neutropenic Infection and Pancytopenia | Up to 6 years
Percentage of Participants Receiving Single-Agent Docetaxel Chemotherapy for Treatment of Relapsed Non-Small Cell Lung Cancer (NSCLC) with an Episode of Neutropenic Sepsis (NS) with an Absolute Neutrophil Count of Less Than 0.5 x 10^9/L | Up to 6 years
Percentage of Participants with Docetaxel-Related Hematological Toxicities, Including Anemia, Thrombocytopenia, Neutropenia, Neutropenic Infection and Pancytopenia | Up to 6 years
Number of Episodes of Neutropenic Sepsis (NS) with an Absolute Neutrophil Count of Less Than 1.0 x 10^9/L | Up to 6 years
Number of Episodes of NS with an Absolute Neutrophil Count of Less Than 0.5 x 10^9/L | Up to 6 years
Number of Episodes of NS Associated with Death Attributable to NS | Up to 6 years
Percentage of Deaths Associated with the Occurrence of an NS Event | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United Kingdom (7):
  - Bristol Haematology and Oncology Centre, Bristol
  - Velindre Cancer Centre, Cardiff
  - Chelsea & Westminster Hospital, London
  - Maidstone Hospital; Kent Oncology Centre, Maidstone
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford
  - Royal Cornwall Hospital, Truro
  - Pinderfields General Hospital; Dept of Haematology, Wakefield